CLINICAL TRIAL: NCT01682395
Title: Best Management of Sigmoid Volvulus: A Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1091
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2015-05

CONDITIONS: Intestinal Volvulus; Colon, Sigmoid
Keywords: Intestinal volvulus; Colon, sigmoid; Anastomosis, surgical; Anastomotic leak; Malawi; Developing Country
MeSH Terms: conditions — Intestinal Volvulus; Anastomotic Leak | interventions — Anastomosis, Surgical; Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- G-SV Resection and colostomy (Active Comparator): Gangrenous sigmoid volvulus patients randomized to undergo resection with colostomy and delayed anastomosis
  Interventions: Procedure: Resection and colostomy
- G-SV Resection and anastomosis (Experimental): Gangrenous sigmoid volvulus subjects randomized to undergo resection and anastomosis
  Interventions: Procedure: Resection and anastomosis
- NG-SV resection and anastomosis (Active Comparator): Nongangrenous sigmoid volvulus subjects randomized to undergo resection and anastomosis
  Interventions: Procedure: Resection and anastomosis
- NG-SV mesosigmoidopexy (Experimental): Nongangrenous sigmoid volvulus subjects randomized to undergo mesosigmoidopexy
  Interventions: Procedure: Mesosigmoidopexy

INTERVENTIONS:
Procedure: Resection and anastomosis — Resection of sigmoid colon with primary anastomosis
  Arms: G-SV Resection and anastomosis; NG-SV resection and anastomosis
Procedure: Resection and colostomy — Resection of sigmoid colon with end colostomy and Hartmann's pouch, followed at a later date by Hartmann's reversal as a second surgical procedure
  Arms: G-SV Resection and colostomy
Procedure: Mesosigmoidopexy — Mesosigmoidopexy--the fixation of the sigmoid colon to lateral abdominal wall with concomitant shortening of the mesosigmoid length.
  Arms: NG-SV mesosigmoidopexy

SUMMARY:
The purpose of this study is to obtain a better understanding of the best management of left-sided colonic emergencies.

DETAILED DESCRIPTION:
Participants: Patients 18 years or older presenting to Kamuzu Central Hospital in Lilongwe Malawi with sigmoid volvulus will be eligible for inclusion.

Procedures (methods): This is a prospective randomized trial. Subjects will be randomized during surgery to receive resection and anastomosis or mesosigmoidopexy (for non-gangrenous sigmoid volvulus), and resection and anastomosis or Hartmann's procedure (for gangrenous sigmoid volvulus).

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of sigmoid volvulus as deemed by the surgeon on duty

Exclusion Criteria:

* pregnancy,
* age under 18 years,
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-Day
  Mortality within 30 days of surgery, as determined by hospital inpatient records, outpatient clinical records and telephone contact (with next-of-kin)per study protocol.

SECONDARY OUTCOMES:
Recurrence of Sigmoid Volvulus | 3 Year
  Recurrence of sigmoid volvulus confirmed radiologically or operatively within 3 years of surgery. This will be determined by hospital inpatient records, outpatient clinical records and telephone contact (with next-of-kin, and if recurrence diagnosed outside of study site contact with the treating physician) per study protocol.
Surgical Site Infection | 30-Day
  Surgical site infections as defined by the Centers for Disease Control within 30 days of surgery.

OTHER OUTCOMES:
Anastomotic Leak | 30-Day
  Communication of the intraluminal and extraluminal space ad defined by clinical presence of a fecal fistula or operative determination of breakdown of the anastomosis within 30 days of surgery. Of note the NG-SV mesosigmoidopexy arm will not be included in this outcome as there is no anastomosis.
Stomal Complications | 3 Year
  Stomal complications (necrosis, pain, skin irritation, retraction, prolapse, stenosis, parastomal herniation, ventral hernia at prior stoma incision) within 3 years of surgery. Of note the G-SV Resection and colostomy arm will be the only arm included in this outcome as none of the other arms include a colostomy.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Samuel, MD, MPH, Principal Investigator — UNC Chapel Hill Department of Surgery
Locations (1):
- Kamuzu Central Hospital, Lilongwe, Malawi

REFERENCES:
- [Background] Raveenthiran V, Madiba TE, Atamanalp SS, De U. Volvulus of the sigmoid colon. Colorectal Dis. 2010 Jul;12(7 Online):e1-17. doi: 10.1111/j.1463-1318.2010.02262.x. Epub 2010 Mar 10. PMID 20236153
- [Background] Akinkuotu A, Samuel JC, Msiska N, Mvula C, Charles AG. The role of the anatomy of the sigmoid colon in developing sigmoid volvulus: a case-control study. Clin Anat. 2011 Jul;24(5):634-7. doi: 10.1002/ca.21131. Epub 2011 Feb 14. PMID 21322064
- [Background] Samuel JC, Msiska N, Muyco AP, Cairns BA, Charles AG. An observational study addressing the anatomic basis of mesosigmoidopexy as a rational treatment of non-gangrenous sigmoid volvulus. Trop Doct. 2012 Jan;42(1):44-5. doi: 10.1258/td.2011.110317. Epub 2011 Dec 19. PMID 22184737
- See also: Related meta-analysis and systematic review registration — http://www.crd.york.ac.uk/prospero/display_record.asp?ID=CRD42012002137